CLINICAL TRIAL: NCT06077669
Title: Multimodal Brain Imaging of the Neural Effects of Methylphenidate in Children and Adolescents With ADHD
Brief Title: Multimodal Brain Imaging of Methylphenidate in Children and Adolescents With ADHD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn in IRB by PI
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00408678
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Methylphenidate - low dose (Experimental): 5 mg of methylphenidate
  Interventions: Drug: Methylphenidate
- Methylphenidate - high dose (Experimental): 10 mg of methylphenidate
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Single oral dose of methylphenidate (5mg or 10 mg)
  Other Names: Ritalin
  Arms: Methylphenidate - high dose; Methylphenidate - low dose
Drug: Placebo — oral placebo
  Arms: Placebo

SUMMARY:
The goal of this proposal is to develop brain imaging tools to measure the effects of methylphenidate in children and adolescents with attention deficit hyperactivity disorder (ADHD). Methylphenidate is an FDA-approved treatment for ADHD. Specifically, the investigators will correlate brain activity during cognitive tasks and brain chemistry with cognitive performance. These measures could help the investigators understand how current ADHD medications work and then could be used to develop novel drugs to treat ADHD in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 18 years
* Diagnosis of ADHD
* A score of at least 3 (mildly ill) on the clinician administered Clinical Global Impressions-Severity (CGI-S)

Exclusion Criteria:

* Currently taking stimulant medications (within one week of first study visit). Patients will not be asked to discontinue any treatments for the purpose of this research study. Subjects will include treatment naïve patients and patients who were previously treated with stimulant medications, but are not currently treated, and meet study criteria.
* Having an adverse reaction to methylphenidate, or other stimulant medication
* Current psychiatric disorder, including bipolar I or II disorder, major depressive, disorder, obsessive-compulsive disorder, autism spectrum disorder, Tourette syndrome, or history of psychosis
* Patient is at risk for clinically significant deterioration due to study protocol, as assessed by primary medical investigator (Dr. Grant)
* Confirmed genetic disorder with cognitive and/or behavioral disturbances
* Active, unstable medical illness that may interfere with cognition or compromises safety of the patient
* History of head trauma with loss of consciousness or any evidence of functional impairment due to, and persisting after, head trauma
* Neurological disorder, mental retardation, intellectual or disability, or other non-ADHD cause of cognitive impairment
* Pregnant or breast-feeding women
* Having a contraindication to MRI, including a pacemaker, defibrillator or other medical implant, other metal objects, or claustrophobia, or for having braces or other metal in the head region (likely to create an artifact on the MRI scans).
* Currently smoking or using controlled or illicit substances, including alcohol.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-16 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
BOLD signal during response inhibition | Approximately 90 minutes after dose
  Blood oxygenation level dependent (BOLD) signal (brain activity during functional magnetic resonance imaging (fMRI), arbitrary units) in the anterior cingulate cortex during response inhibition.
BOLD signal during working memory | Approximately 90 minutes after dose
  BOLD signal (brain activity during fMRI, arbitrary units) in the frontal cortex during working memory
Glutamate level in the anterior cingulate cortex | Approximately 2 hours after dose
  Glutamate level (measured by magnetic resonance spectroscopy (MRS), institutional units) in the anterior cingulate cortex (ACC).
Glutamate level in the dorsolateral prefrontal cortex | Approximately 2 hours after dose
  Glutamate level (measured by MRS, institutional units) in the dorsolateral prefrontal cortex
Cognitive performance as assessed by the Flanker performance task | Approximately 3 hours after dose
  NIH Toolbox Cognitive Battery Flanker task, score range 0 to 20, higher score is better performance
Working memory performance | Approximately 3 hours after dose
  NIH Toolbox Cognitive Battery working memory task (list sorting), score range 0 to 26, higher score is better performance

SECONDARY OUTCOMES:
ADHD as assessed by the Connors 3 | At each study visit, approximately 3 hours after dose
  Connors 3rd edition ADHD assessment, lower score means less symptoms, typical scores are 40 to 59, above 65 is an elevated score (meaning more concerns than are typically reported)
NIH Toolbox Cognitive Battery | Approximately 3 hours after dose
  Cognition Fluid Composite, Cognition Crystallized Composite, Cognition Total Composite Score, and other individual test scores
Methylphenidate plasma levels | Approximately 90 min and 150 min after dose
  Methylphenidate plasma levels will be drawn before and after brain imaging on each visit

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bigos, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be deposited in the National Institute of Mental Health Data Archive (NDA) will be collected for each subject. All raw and processed phenotypic data (clinical, cognitive, imaging) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be deposited at 12 months after the start of recruitment, and every 6 months following